CLINICAL TRIAL: NCT03224494
Title: Evaluation of Visceral Bowel Sensitivity Threshold in Irritable Bowel Syndrome Patients Versus in Healthy Controls Using the Novel Rapid Barostat Bag
Brief Title: Evaluation of Bowel Sensitivity Threshold in IBS Patients Versus in Healthy Controls Using the Novel Rapid Barostat Bag
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Stephen Vanner, Professor, Queen's University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6021016
Record Dates: First submitted 2017-07-07; First posted 2017-07-21 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Irritable Bowel Syndrome; Visceral Hypersensitivity
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBS Patients (Other): Patients 18 years or older with a diagnosis of irritable bowel symptom, as per Rome IV criteria. The diagnosis is established by the patient's gastroenterologist. Please see inclusion and exclusion section for more details.
  They will undergo Rapid Barostat Bag testing, and they will answer the IBS severity scoring system questionnaire (IBS-SSS) and HAD scale questionnaire.
  Interventions: Device: Rapid Barostat Bag; Other: IBS severity scoring system questionnaire (IBS-SSS); Other: HAD scale questionnaire
- Healthy Controls (Other): Patients 18 years of age without IBS or other colo-rectal symptoms or pathology seen for other issues in the general GI clinic.
  They will undergo Rapid Barostat Bag testing, and they will answer the IBS severity scoring system questionnaire (IBS-SSS) and HAD scale questionnaire.
  Interventions: Device: Rapid Barostat Bag; Other: IBS severity scoring system questionnaire (IBS-SSS); Other: HAD scale questionnaire

INTERVENTIONS:
Device: Rapid Barostat Bag — Both healthy controls (n= 100) and IBS patients (n=100) will undergo anorectal studies using a Rapid barostat bag catheter.
Other: IBS severity scoring system questionnaire (IBS-SSS) — We will correlate the changes to IBS symptoms using the IBS severity scoring system questionnaire (IBS-SSS). The questionnaire will be administered twice for IBS patients who have consented to return for a second study visit, at each of the two RBB studies.
Other: HAD scale questionnaire — It is a validated anxiety and depression questionnaire

SUMMARY:
BACKGROUND & AIMS: Bowel hypersensitivity (lower threshold for discomfort in response to distention of a balloon in the rectum compared to healthy controls) is a key documented feature in Irritable Bowel Syndrome (IBS) mechanistic studies. The use of the barostat catheter to assess bowel hypersensitivity has been well documented in research settings, but it's use is time consuming which makes it unpractical for routine clinical practice (test time up to 60 minutes). The Rapid Barostat Bag is a novel device used to obtain a rapid and simple assessment of the rectal function, which has received approval for use by Health Canada. Although its safety and use has been validated in healthy controls, RBB use has never been reported in a cohort of IBS patients. The aim of this study is to 1) evaluate bowel sensitivity in IBS patients, compared with healthy controls and 2) determine whether the sensory threshold predicts response to standard of care interventions such as diet or medications.

METHODS: This is a prospective controlled study. All participants will undergo RBB testing and will answer a questionnaire related to bowel symptoms (IBS-SSS - IBS Severity Scoring System) and a questionnaire related to anxiety/depression (HADS - Hospital and Anxiety and Depression Scale).

HYPOTHESIS: The investigators hypothesize that IBS patients will display lower bowel sensitivity thresholds than healthy controls, using the RBB device. Furthermore, we predict that those with a low sensory threshold (i.e. visceral hypersensitivity) are most likely to respond to interventions that decrease bowel distention (e.g. low FODMAP diet) or the medication linaclotide that is reported to decrease pain signaling.

DETAILED DESCRIPTION:
IBS is a clinical entity characterized by abdominal pain and altered bowel movements. About 20% of the western population is affected by IBS. Abnormal perception of visceral stimuli plays a paramount role in the pathogenesis of IBS related abdominal pain. Moreover, sensitization (modulation of intracellular mechanisms leading to exaggerated action potential discharge in response to a given stimulus) of nociceptive dorsal root ganglia (DRG) neurons by tissue mediators is a fundamental mechanism underlying abnormal pain signaling. Clinical management of IBS has consisted primarily of symptomatic management of the altered bowel movement pattern. Although these can also afford improvement in abdominal pain, pharmacotherapy directly targeting bowel hypersensitivity are limited. Tri-cyclic antidepressants have been used in small doses in selected IBS patients who have not responded to first line therapy, but anti-cholinergic side effects have limited their use. The low FODMAP diet is well described therapeutic intervention which also targets bowel hypersensitivity, and about 70% of patients respond to this intervention. However, predictors of response to the various IBS therapies are lacking, and treatment decisions are often made on a "trial and error" fashion.

Assessment of bowel sensitivity has been reported using a barostat (an elastic balloon inflated manually by a syringe until rectal sensations are reported). Unfortunately, barostat device use has not been practical because considerable time is required to carry out the studies (up to 60 min). As such, barostat studies have been used mainly in research settings.

The rapid barostat bag (RBB) is a novel handheld barostat device. It is quick and simple to use, and its polyethylene bag provides superior volume measurements than the elastic balloons currently in use. This test could ultimately provide a bedside measure in the clinic of patients and identify those who are hypersensitive and thus more likely to respond to therapies targeting this sensory disorder. Data on validation of the RBB method against the standard barostat system has been published, using healthy volunteers. However, no studies evaluating the use of the RBB to assess bowel visceral sensitivity have been published to date.

Thus, there are 2 aims to this study:

Aim 1. To evaluate bowel sensitivity in IBS patients, compared with healthy controls.

Aim 2. To determine whether sensory thresholds measured in clinic at the time of the initial physical examination correlate with standard of care interventions, such as a low FODMAP diet or medication such as linaclotide.

This new knowledge will afford the opportunity to gain new insights into the bowel hypersensitivity which characterizes IBS. The overall goal of this study will be to assess if IBS-mediated bowel hypersensitivity as assessed by the RBB can serve as predictor of response to IBS pharmacotherapy.

Both healthy controls (n= 100) and IBS patients (n=100) will undergo anorectal studies using a Rapid barostat bag catheter. To test for stability of the response over time, IBS patients will be given the option of returning in one month time so these studies can be repeated. These studies will measure rectal perception to balloon inflation. The investigators will correlate the changes to IBS symptoms using the IBS severity scoring system questionnaire (IBS-SSS). The questionnaire will be administered twice for IBS patients who have consented to return for a second study visit, at each of the two RBB studies. The patients will also complete a validated anxiety and depression questionnaire (HAD scale). The symptom questionnaires will also be administered to the healthy controls, to prove that they indeed do not have symptoms of IBS. The Rapid Barostat Bag (Mui Scientific, Mississauga) will be used for these studies. It has been approved for clinical use by Health Canada. It is a computer driven volume displacement device. The device measures pressures and volumes (sampling rate 1-2mL/second) and is connected to a device that monitors sensations as 0= no pain,1=sensation, 2=urge, 3=discomfort.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with IBS by their treating gastroenterologist, according to the Rome IV criteria. According to Rome IV criteria, IBS is defined as:

   recurrent abdominal pain, on average, at least one day per week in the last three months, associated with 2 or more of the following:
   1. pain is related to defecation
   2. associated with a change in stool frequency
   3. associated with a change in stool form.
2. Irritable Bowel syndrome patients will be recruited from the GI motility clinic and general GI clinic at Hotel Dieu Hospital.
3. Healthy controls will be recruited from the GI clinics. These are patients coming for evaluation for non-colonic symptoms such as colon screening, gastroesophageal reflux disease, or liver disease.

Exclusion Criteria:

1. patients under the age of 18;
2. a recent change in IBS treatment regimen or patients taking analgesics, which may affect bowel sensitivity (this includes the FODMAP diet)
3. pregnant patients, as there may be a small risk of inducing labor with the barostat probe
4. patients who have had previous colorectal surgery as it may bowel sensitivity
5. healthy controls who are experiencing bowel symptoms
6. known significant anorectal pathology (eg. fistulae, abscess, stricture, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-08-10 (Actual); Primary Completion 2019-07-15 (Estimated); Study Completion 2019-07-15 (Estimated)

PRIMARY OUTCOMES:
Bowel sensory threshold | A second visit to record sensory threshold a second time may be obtained up to 52 weeks after the first visit.
  Sensory thresholds are obtained via rapid barostat bag measurements, and are expressed in millilitres.

SECONDARY OUTCOMES:
IBS-SSS Questionnaire | At first visit, and during a second visit. A second visit may be obtained up to 52 weeks after the first visit.
  This is a validated symptom questionnaire pertaining to irritable bowel syndrome symptoms.
HADS scale questionnaire | At first visit, and during a second visit. A second visit may be obtained up to 52 weeks after the first visit.
  This is a validated questionnaire pertaining to psychological parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Vanner, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston Health Sciences Centre - HDH site, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There will be no sharing of individual participation data with other researchers

REFERENCES:
- [Background] Sauter M, Heinrich H, Fox M, Misselwitz B, Halama M, Schwizer W, Fried M, Fruehauf H. Toward more accurate measurements of anorectal motor and sensory function in routine clinical practice: validation of high-resolution anorectal manometry and Rapid Barostat Bag measurements of rectal function. Neurogastroenterol Motil. 2014 May;26(5):685-95. doi: 10.1111/nmo.12317. Epub 2014 Feb 12. PMID 24517865
- [Background] Halmos EP, Power VA, Shepherd SJ, Gibson PR, Muir JG. A diet low in FODMAPs reduces symptoms of irritable bowel syndrome. Gastroenterology. 2014 Jan;146(1):67-75.e5. doi: 10.1053/j.gastro.2013.09.046. Epub 2013 Sep 25. PMID 24076059